CLINICAL TRIAL: NCT06859762
Title: A Phase 1, Multicenter, Open-Label, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of YL217 in Patients With Advanced Solid Tumors
Brief Title: A First-in-Human Study of YL217 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL217-INT-101-01
Record Dates: First submitted 2025-02-18; First posted 2025-03-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: A Phase 1, Multicenter, Open-Label, First-in-Human Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 2: The backfill stage of YL217 (Experimental): Patients will be enrolled at one or more dose levels that do not exceed the dose that is deemed safe and tolerable in dose escalation. Then several dose levels will be selected as the recommended dose for expansion (RDE).
  Interventions: Drug: YL217
- Part 1: Dose-Escalation Part (Experimental): Participants will receive escalating doses of YL217 until doses for optimization are determined
  Interventions: Drug: YL217
- Part 3: Dose-Expansion Part (Experimental): Upon completion of Part 1 and Part 2 with determination of MTD/RDE(s), the dose-expansion part will be conducted to further support the RP2D selection.
  Interventions: Drug: YL217

INTERVENTIONS:
Drug: YL217 — Patients will be treated with YL217 intravenous(IV)infusion.
  Arms: Part 1: Dose-Escalation Part
Drug: YL217 — Patients will be treated with YL217 intravenous(IV)infusion.
  Arms: Part 3: Dose-Expansion Part
Drug: YL217 — Patients will be treated with YL217 intravenous(IV)infusion.
  Arms: Part 2: The backfill stage of YL217

SUMMARY:
A Phase 1 First-in-Human study of YL217 in Patients with Advanced Solid Tumors

DETAILED DESCRIPTION:
YL217 is an antibody-drug conjugate (ADC) that targets CDH17 (Cadherin-17) protein and is being developed for the treatment of cancer. YL217 is comprised of three components: 1) YL217-mAb, a CDH17-targeting recombinant humanized immunoglobulin G1 (IgG1) monoclonal antibody, 2) YL0010014, a topoisomerase I inhibitor, and 3) an enzymatically cleavable methylsulfonyl pyrimidine tripeptide drug linker.

The in vivo anti-tumor efficacy of YL217 was evaluated in immune-deficient mice bearing human colorectal cancer, gastric cancer and patient derived colorectal cancer xenograft tumors. The results indicated that YL217 was well tolerated, and YL217 suppressed growth of established human tumors in a dose-dependent manner in cancer cells or patient derived xenograft models.

Therefore, in order to meet the huge unmet medical needs in the field of gastrointestinal cancer treatment, it is planned to conduct the first human phase I clinical study of YL217 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Informed of the study before the start of the study and voluntarily sign their name and date in the ICF
* Able and willing to comply with protocol visits and procedures
* Age≥ 18 years
* ECOG PS of 0 or 1
* Tumor types as below:

For Part 1 and Part 2: Pathologically confirmed diagnosis of an advanced solid tumor.

For Part 3 (Histologically or cytologically confirmed diagnosis+ locally advanced unresectable or metastatic disease)

* Adequate organ and bone marrow function.
* Have at least 1 extracranial measurable tumor lesion.
* Adequate archival formalin-fixed paraffin embedded （FFPE） tissue from prior biopsy.

Exclusion Criteria:

* Prior treatment with an agent targeting CDH17
* Prior discontinuation of a topoisomerase I inhibitor due to treatment-related toxicities.
* Have received an ADC consisting of a topoisomerase I inhibitor.
* Concurrent enrollment in another clinical study, unless it is an observational clinical study.
* Inadequate washout period for prior anticancer treatment before the first dose of study drug
* Undergone major surgery within 4 weeks before the first dose of study drug or expect major surgery during the study.
* Received long term systemic steroids or other immunosuppressive therapy within 2 weeks before the first dose of study drug.
* Received any live vaccine within 4 weeks before the first dose of study drug or intend to receive a live vaccine during the study.
* Diagnosis or evidence of spinal cord compression or leptomeningeal carcinomatosis.
* Uncontrolled or clinically significant cardiovascular and cerebrovascular diseases.
* A history of non-infectious interstitial lung disease (ILD)/pneumonitis that requires steroids, current active ILD/pneumonitis.
* Have clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses.
* Uncontrolled third-space fluid that requires repeated drainage.
* Digestive system disease that may cause bleeding, perforation, jaundice, gastrointestinal obstruction.
* An active tuberculosis based on medical history.
* Known human immunodeficiency virus (HIV) infection.
* Active hepatitis C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Nature and frequency of dose-limiting toxicity(DLT) | Up to approximately 3 years
  The purpose of DLT is to find maximum tolerated dose (MTD).
Nature and frequency of adverse events (AEs) with severity | Up to approximately 3 years
  Nature and frequency of AEs with severity is aim to evaluate the safety of YL217.
objective response rate (ORR) | Up to approximately 3 years
  ORR: defined as the proportion of patients who achieved a best overall response of complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Eastern Cooperative Oncology Group performance status (ECOG PS) | Up to approximately 3 years
  Deterioration of Eastern Cooperative Oncology Group performance status (ECOG PS)
To evaluate safety endpoint of peripheral oxygen saturation (SpO2) | Up to approximately 3 years
Characterize Pharmacokinetics(PK) parameter AUC | Up to approximately 3 years
  The area under curve: AUC is the total amount of YL217 in bloodstream after drug administration.
Characterize Pharmacokinetics(PK) parameter Cmax | Up to approximately 3 years
  Maximum concentration：The highest measured concentration of YL217 in the bloodstream.
Characterize Pharmacokinetics(PK) parameter Ctrough | Up to approximately 3 years
  Trough concentration
Characterize Pharmacokinetics(PK) parameter Tmax | Up to approximately 3 years
  Time to maximum observed concentration
Characterize Pharmacokinetics(PK) parameter CL | Up to approximately 3 years
  Clearance： defined as the amount of drug removed from the bloodstream by the body per unit of time.
Characterize Pharmacokinetics(PK) parameter Vd | Up to approximately 3 years
  volume of distribution
Characterize Pharmacokinetics(PK) parameter t1/2 | Up to approximately 3 years
  Half-life time：defined as the time it takes for the concentration of the drug in plasma or serum to be reduced by 50%.
Immunogenicity endpoint: Incidence of anti-YL217 antibody (ADAs). | Up to approximately 3 years
  The presence of ADAs in patients treated with YL217 will be assessed to evaluate immunogenicity.
Disease control rate (DCR) | Up to approximately 3 years
  DCR: defined as the proportion of patients who achieved a best overall response of complete response (CR), partial response (PR) or stable disease (SD).
Duration of response (DoR) | Up to approximately 3 years
  DoR: defined as the time interval from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of progressive disease (PD).
Time to response (TTR) | Up to approximately 3 years
  TTR: defined as the time interval from the date of the first dose of study drug to the date of the first documentation of objective response (CR or PR).
Depth of response (DpR) | Up to approximately 3 years
  DpR: defined as the proportion of target lesion shrinkage from baseline to maximum tumor size.
Progression-free survival (PFS) | Up to approximately 3 years
  PFS: defined as the time interval from the date of the first dose of study drug to the date of first documentation of PD or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to approximately 3 years
  OS: defined as the time interval from the date of the first dose of study drug to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (13):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - The University of Kansas Cancer Center (KUCC), Kansas City, Kansas
  - University of Maryland Medical Center-Greenebaum Cancer Ctr - Medical Oncology, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Columbia University Irving Medical Center, New York, New York
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - UT Health San Antonio - Mays Cancer Center, San Antonio, Texas
  - University of Wisconsin Health - UW Carbone Cancer Center, Madison, Wisconsin
- China (6):
  - Peking Union Medical College Hospital, Beijing, Bejing
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No